CLINICAL TRIAL: NCT07022275
Title: Safety Evaluation of THC-Free Hemp Protein Isolate
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Natural Medicine (Other)
Responsible Party: Principal Investigator, Brice Thompson, Clinical Investigator, National University of Natural Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BT10124
Record Dates: First submitted 2025-05-30; First posted 2025-06-15 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-05

CONDITIONS: Tolerability of Hemp Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hemp Protein (Experimental): Healthy adults consuming 20 grams of Hemp Protein Powder twice a day for 30 days
  Interventions: Dietary Supplement: Hemp protein powder

INTERVENTIONS:
Dietary Supplement: Hemp protein powder — Agoge Universal Hemp Protein Powder - A certified cannabinoid-free hemp protein powder.

SUMMARY:
The goal of this clinical trial is to evaluate the safety and tolerability of a THC-free hemp protein supplement in healthy adult volunteers aged 18-65 years who do not use cannabis or hemp-derived products. The main questions this study aims to answer are:

Does twice-daily consumption of 20 grams of Agoge Hemp Protein Powder for 30 days result in detectable levels of THC-COOH, the primary metabolite of THC, in urine samples? Is the supplement well tolerated, and does it affect common clinical safety markers (e.g., liver and kidney function, inflammatory markers)?

This is a single-arm study with no comparison group. All participants will:

* Consume 20 grams of the hemp protein supplement twice daily for 30 days
* Provide blood and urine samples at baseline and Day 30
* Complete weekly surveys assessing adherence, tolerability, and adverse events

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years.
* Able and willing to provide informed consent.
* In good general health as determined by medical history and screening.
* No cannabis or hemp product use within the past 90 days and willingness to avoid consuming other hemp-based or cannabinoid-containing products during the study period.
* Willing to take 20 grams of hemp protein powder, twice a day, for 30 days, complete two blood draws, provide two urine samples, and fill out weekly surveys.

Exclusion Criteria:

* Positive THC-COOH baseline urine test.
* Regular use of any medications that could interfere with THC metabolism.
* History of substance abuse or dependence within the past year.
* Individuals who are pregnant, lactating, or planning a pregnancy within the next 30 days.
* Known allergy or hypersensitivity to cannabis, hemp, or any component of the study product.
* Participants with chronic liver, kidney, or severe cardiovascular disease.
* Participants with dietary restrictions that may prevent them from consuming the study product.
* Current or recent participation in another research study within 14 days of screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-09-25 (Estimated); Study Completion 2025-09-25 (Estimated)

PRIMARY OUTCOMES:
Presence of THC-COOH in Urine | 30 days
  To determine whether THC-COOH, the primary metabolite of THC, is detectable in participants' urine after 30 days of consuming 40 grams of Agoge Hemp Protein Powder.

SECONDARY OUTCOMES:
Number of participants who develop ≥ 1 new clinically-significant laboratory abnormality (hematology, hepatic, or renal) between baseline and day 30. | Baseline (Day 0) and End of Study (Day 30)
  A 'clinically-significant laboratory abnormality' is defined as any value judged by the principal investigator to be new-onset or ≥ 1 severity grade and rated as at least 'possibly related' to the study product, using CTCAE v5.0 grading where available. CBC - hemoglobin, hematocrit, WBC, or platelet count that shifts from normal at baseline to below/above reference limits by ≥ 1 CTCAE grade. Hepatic Panel - AST or ALT rises to > 2 x upper limit of normal (ULN). Renal Panel - estimated glomerular filtration rate (eGFR) falls to < 60 mL/min/1.73 m^2 or decreases by ≥ 25% from baseline; blood-urea-nitrogen-to-creatinine ratio (BUN:Cr) rises above 20:1 if previously normal. Venous blood is drawn at day 0 and day 30 for CBC, CMP, and calculated eGFR. Results are entered into REDCap, reviewed by a clinician, and coded for relatedness and severity. The study will report n/N (%) of participants meeting any abnormality criterion.
Number of participants who experience ≥ 1 treatment-emergent adverse event related to the product | 30 days - Participants complete the REDCap Survey on days 7, 14, 21, and 28
  Any self-reported adverse event (AE) deemed at least "possibly related" to the study product. Data collection will occur through a 7-item symptom questionnaire through a REDCap Survey querying about nausea, headache, dizziness, fatigue, skin reactions, gastrointestinal issues, or any other unsolicited symptoms. If any symptom is reported, study staff complete a standardized spontaneous AE reporting form. Each AE is graded for severity (mild, moderate, severe) and relatedness (unrelated, possibly, probably, or definitely) by study staff. The count and proportion of participants experiencing ≥ product-related AE over the 30-day intervention will be reported (n/N [%])

CONTACTS AND LOCATIONS:
Locations (1):
- Helfgott Research Institute, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No